CLINICAL TRIAL: NCT04275362
Title: Gait Analysis of a Lateral-Pivot Design Total Knee Replacement
Status: Recruiting | Type: Observational
Sponsor: More Foundation (Other)
Collaborators: Encore Medical, L.P. (Industry)
Responsible Party: Sponsor
Other Study IDs: 4015
Record Dates: First submitted 2020-02-12; First posted 2020-02-19 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Total knee arthroplasty; Lateral pivot
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (6):
- DJO subjects for surgical technique: Subjects who meet the inclusion criteria and receive a DJO Empowr total knee replacement but will not participate in motion data collection
  Interventions: Device: DJO Empowr PS Knee System
- DJO subjects for data collection: Subjects who meet the inclusion criteria and consent to be in the study will receive a DJO Empowr total knee replacement and participate in motion data collections at pre-op, and 6 and 12 months post-op. Subjects will also participate in pre-op, 6 month, 1 year, 2 year, 5 year, and 10 year post-op clinical data collections
  Interventions: Device: DJO Empowr PS Knee System
- Prospective control subjects: Healthy age matched subjects who did not have any knee osteoarthritis and participated in motion data collections.
  Interventions: Device: Control
- Stryker TKA subjects: Subjects who met the inclusion criteria and consented to be in a study whereby they received a Stryker Triathlon total knee replacement and participated in motion analysis pre-surgery and 6 and 12 months post-surgery.
  Interventions: Device: Stryker Triathlon Total Knee System
- Biomet TKA subjects: Subjects who met the inclusion criteria and consented to be in a study whereby they received a Biomet Vanguard total knee replacement and participated in motion analysis pre-surgery and 12 months post-surgery.
  Interventions: Device: Biomet Vanguard Complete Knee System
- Retrospective control subjects: Healthy age matched subjects who did not have any knee osteoarthritis and participated in motion data collections.
  Interventions: Device: Control

INTERVENTIONS:
Device: DJO Empowr PS Knee System — Patients will receive a DJO Empowr PS Knee System total knee replacement
  Groups: DJO subjects for data collection; DJO subjects for surgical technique
Device: Stryker Triathlon Total Knee System — Patients received a Stryker Triathlon Total Knee System total knee replacement
  Groups: Stryker TKA subjects
Device: Biomet Vanguard Complete Knee System — Patients received a Biomet Vanguard Complete Knee System total knee replacement
  Groups: Biomet TKA subjects
Device: Control — No total knee replacement
  Groups: Prospective control subjects; Retrospective control subjects

SUMMARY:
Previous motion analysis studies have demonstrated excellent ability to distinguish subtle differences in gait between normal subjects and those suffering from arthritis. With proper techniques and analysis differences between osteoarthritis patient groups can be distinguished. Previous research has indicated that subjects who received a single-radius design total knee replacement have superior gait performance that those who received a multi-radius design total knee replacement. The DJO Global Empowr PS Knee System is a single-radius lateral pivot design. This design should achieve reproducible more natural knee function and improved patient outcomes and satisfaction. A motion analysis laboratory will be used to collect gait data from patients who are going to receive a Empowr PS knee device and also from age-matched control subjects. These data will be compared with data previously collected from patients who received Stryker Triathlon devices, Biomet Vanguard devices and age-matched healthy control subjects.

DETAILED DESCRIPTION:
Thirty subjects who are scheduled to receive an Empowr PS Total Knee Replacement device will be consented to be in the prospective component of the study. Twenty of these patients will participate in motion data collection. These patients will all be scheduled to undergo primary total knee replacement using the Empowr device. All surgeries will be performed using computer navigation. Patients will receive standardized physical therapy to insure consistency of rehab protocols and discharge from physical therapy criteria. Specifically, patients will be monitored for visit compliance, Timed Up and Go (TUG) test in seconds, AROM in degrees, and walking un-aided.

Data were previously collected preoperatively, at 6 months and 1 year post-operatively for 16 patients who received a Stryker Triathlon total knee replacement and preoperatively and 1 year post-op for 16 patients who received a Biomet Vanguard total knee replacement. Data were also previously collected for 20 age matched healthy controls subjects. Data will be collected for an additional 20 control subjects. Knee Society Score (KSS) and Knee Injury and Osteoarthritis Outcome Score (KOOS) will be collected at pre-op, 6 months, 1 year, and 2 years post-op. Gait analysis data will include kinetic, kinematic, temporal spatial, and electromyographic (EMG) data throughout the gait cycle for both research subjects and controls. Reflective markers will be placed on subject's anatomical landmarks, and ten surface EMG electrodes placed according to published standards (8). Subjects will walk at a self-selected speed down a runway embedded with force plates while 10 Eagle-4 digital infrared cameras record their movement. In addition to the level surface walking, additional data on more complex activities of daily living will be collected for potential future analysis. This would include: sit-to-stand, balance, and stair-climbing measurements also using the force plates, camera system and EMG data collection.

ELIGIBILITY:
Inclusion Criteria:

Controls:

1. At least 50 years of age.
2. Subjects who provide signed and IRB approved informed consent for gait analysis data collection

Retrospective subjects:

1. Subjects who had primary total knee replacement with either Stryker Triathlon Total Knee System or Biomet Vanguard Complete Knee System.
2. Subjects at least 50 years of age at the time of the surgery.
3. Subjects who previously provided signed and informed consent for gait analysis data collection under approval of the Sun Health Institutional Review Board
4. Cases that followed product labeling.

Prospective subjects:

1. Subjects who are eligible for DJO Global's Empowr total knee replacement.
2. Subjects at least 50 years of age at the time of the surgery.
3. Subjects who are willing to provide signed and IRB approved informed consent for gait analysis data collection.
4. Cases that followed product labeling.

Exclusion Criteria:

Controls:

1. Controls with any musculoskeletal injury or disorder.
2. Controls that are pregnant or planning on becoming pregnant.
3. Controls with a BMI>40

Retrospective subjects:

1. Subjects with inflammatory arthritis or psoriatic arthritis at the time of surgery.
2. Subjects that are pregnant or planning on becoming pregnant.
3. Subjects with a BMI>40
4. Subjects who had an active infection or suspected latent infection in or about the joint at the time of surgery.
5. Subjects whose bone stock was compromised by disease, infection or prior implantation which could not provide adequate support and/or fixation of the prosthesis.
6. Subjects who had any mental or neuromuscular disorders which created an unacceptable risk of prosthesis instability, prosthesis fixation failure, or complication in postoperative care.
7. Subjects with severe instability of the knee joint secondary to the absence of collateral ligament integrity and function.

Prospective subjects:

1. Subjects with inflammatory arthritis or psoriatic arthritis at the time of surgery.
2. Subjects that are pregnant or planning on becoming pregnant.
3. Subjects with a BMI>40
4. Subjects who had an active infection or suspected latent infection in or about the joint at the time of surgery.
5. Subjects whose bone stock was compromised by disease, infection or prior implantation which could not provide adequate support and/or fixation of the prosthesis.
6. Subjects who had any mental or neuromuscular disorders which created an unacceptable risk of prosthesis instability, prosthesis fixation failure, or complication in postoperative care.
7. Subjects with severe instability of the knee joint secondary to the absence of collateral ligament integrity and function.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 4 groups: 1) Healthy age matched controls, 2) Retrospective subjects who have previously received either a Stryker Triathlon TKA or a Biomet Vanguard TKA and participated in IRB approved gait analysis at pre-op, 6 month, and 12 month post-op time points
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2017-02-02 (Actual); Primary Completion 2023-04-02 (Estimated); Study Completion 2029-01-02 (Estimated)

PRIMARY OUTCOMES:
Knee flexion angle during swing | Pre-op
  Compare maximum knee flexion angle in degrees during swing between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Knee flexion angle during swing | 6 months post-op
  Compare maximum knee flexion angle in degrees during swing between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
Knee flexion angle during swing | 12 months post-op
  Compare maximum knee flexion angle in degrees during swing between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Knee flexion angle during stance | pre-op
  Compare maximum knee flexion angle in degrees during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Knee flexion angle during stance | 6 months post-op
  Compare maximum knee flexion angle in degrees during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
Knee flexion angle during stance | 12 months post-op
  Compare maximum knee flexion angle in degrees during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Knee adduction angle during stance | pre-op
  Compare maximum knee adduction angle in degrees during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Knee adduction angle during stance | 6 months post-op
  Compare maximum knee adduction angle in degrees during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
Knee adduction angle during stance | 12 months post-op
  Compare maximum knee adduction angle in degrees during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.knee replacement (DJO Empowr) and single-radius (Triathlon, Stryker) and multi-radius (Vanguard, Zimmer Biomet) knee replacements.
Knee flexion moment | pre-op
  Compare maximum knee flexion moment normalised to subject body weight (N-m/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Knee flexion moment | 6 months post-op
  Compare maximum knee flexion moment normalised to subject body weight (N-m/kg) during stance between between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
Knee flexion moment | 12 months post-op
  Compare maximum knee flexion moment normalised to subject body weight (N-m/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Knee adduction moment | Pre-op
  Compare maximum knee adduction moment normalised to subject body weight (N-m/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Knee adduction moment | 6 months post-op
  Compare maximum knee adduction moment normalised to subject body weight (N-m/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), oe a single-radius (Triathlon, Stryker) knee replacement.
Knee adduction moment | 12 months post-op
  Compare maximum knee adduction moment normalised to subject body weight (N-m/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Knee power | Pre-op
  Compare maximum knee power in the sagittal plane normalised to subject body weight (W/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Knee power | 6 month post-op
  Compare maximum knee power in the sagittal plane normalised to subject body weight (W/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
Knee power | 12 month post-op
  Compare maximum knee power in the sagittal plane normalised to subject body weight (W/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Vertical GRF | pre-op
  Compare maximum vertical ground reaction force normalised to subject body weight (unitless) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Vertical GRF | 6 months post-op
  Compare maximum vertical ground reaction force normalised to subject body weight (unitless) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
Vertical GRF | 12 month post-op
  Compare maximum vertical ground reaction force normalised to subject body weight (unitless) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
AP GRF | Pre-op
  Compare maximum anterior-posterior ground reaction force normalised to subject body weight (unitless) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
AP GRF | 6 months post-op
  Compare maximum anterior-posterior ground reaction force normalised to subject body weight (unitless) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
AP GRF | 12 months post-op
  Compare maximum anterior-posterior ground reaction force normalised to subject body weight (unitless) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
ML GRF | pre-op
  Compare maximum medial-lateral ground reaction force normalised to subject body weight (unitless) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
ML GRF | 6 months post-op
  Compare maximum anterior-posterior ground reaction force normalised to subject body weight (unitless) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
ML GRF | 12 months post-op
  Compare maximum anterior-posterior ground reaction force normalised to subject body weight (unitless) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.

SECONDARY OUTCOMES:
Ankle dorsiflexion angle during swing | Pre-op
  Compare maximum ankle dorsiflexion angle in degrees during swing between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Ankle dorsiflexion angle during swing | 6 months post-op
  Compare maximum ankle dorsiflexion angle in degrees during swing between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
Ankle dorsiflexion angle during swing | 12 months post-op
  Compare maximum ankle dorsiflexion angle in degrees during swing between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Ankle plantarflexion angle during stance | pre-op
  Compare maximum ankle plantarflexion angle in degrees during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Ankle plantarflexion angle during stance | 6 months post-op
  Compare maximum ankle plantarflexion angle in degrees during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
Ankle plantarflexion angle during stance | 12 months post-op
  Compare maximum ankle plantarflexion angle in degrees during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Ankle plantarflexion moment during stance | pre-op
  Compare maximum ankle plantarflexion moment normalised to subject body weight (N-m/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Ankle plantarflexion moment during stance | 6 months post-op
  Compare maximum ankle plantarflexion moment normalised to subject body weight (N-m/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
Ankle plantarflexion moment during stance | 12 months post-op
  Compare maximum ankle plantarflexion moment normalised to subject body weight (N-m/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Ankle power | Pre-op
  Compare maximum ankle power in the sagittal plane normalised to subject body weight (W/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Ankle power | 6 months post-op
  Compare maximum ankle power in the sagittal plane normalised to subject body weight (W/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
Ankle power | 12 months post-op
  Compare maximum ankle power in the sagittal plane normalised to subject body weight (W/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Hip flexion maximum during swing | Pre-op
  Compare hip flexion angle in degrees during swing between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Hip flexion during swing | 6 months post-op
  Compare maximum hip flexion angle in degrees during swing between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
Hip flexion during swing | 12 months post-op
  Compare maximum hip flexion angle in degrees during swing between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Hip extension during stance | Pre-op
  Compare maximum hip extension angle in degrees during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Hip extension during stance | 6 months post-op
  Compare maximum hip extension angle in degrees during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Hip extension during stance | 12 months post-op
  Compare maximum hip extension angle in degrees during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Hip flexion moment during stance | Pre-op
  Compare maximum hip flexion moment normalised to subject body weight (N-m/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Hip flexion moment during stance | 6 months post-op
  Compare maximum hip flexion moment normalised to subject body weight (N-m/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
Hip flexion moment during stance | 12 months post-op
  Compare maximum hip flexion moment normalised to subject body weight (N-m/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Hip power | Pre-op
  Compare maximum hip power in the sagittal plane normalised to subject body weight (W/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
Hip power | 6 months post-op
  Compare maximum hip power in the sagittal plane normalised to subject body weight (W/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
Hip power | 12 months post-op
  Compare maximum hip power in the sagittal plane normalised to subject body weight (W/kg) during stance between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
KSS | Pre-op
  Compare Knee Society Score between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
KSS | 6 months post-op
  Compare Knee Society Score between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
KSS | 12 months post-op
  Compare Knee Society Score between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
LEAS | Pre-op
  Compare Lower Extremity Activity Score between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.
LEAS | 6 months post-op
  Compare Lower Extremity Activity Score between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), or a single-radius (Triathlon, Stryker) knee replacement.
LEAS | 12 months post-op
  Compare Lower Extremity Activity Score between healthy controls, and subjects with a dual pivot design total knee replacement (DJO Empowr), a single-radius (Triathlon, Stryker) knee replacement or a multi-radius (Vanguard, Zimmer Biomet) knee replacement.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Siverhus, MD, Principal Investigator — The CORE Institute
Locations (1):
- MORE Foundation, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No